CLINICAL TRIAL: NCT07052461
Title: Association of Microcirculation, Vexus Score and Femoral Vein Doppler in Patients on the ICU After Non-emergency Cardiac Surgery
Acronym: VeMic
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00579; am24Siegemund
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Microcirculatory Diffusion; Microcirculatory Convection Capacity; Venous Congestion; Postoperative Cardiac Surgery; Fluid Management; Haemodynamic Coherence
Keywords: vexus score; femoral vein doppler; intensive care unit
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the VeMic study is to explore if venous congestion is linked with microcirculatory impairment in elective cardiac surgery patients in the postoperative ICU stay.

DETAILED DESCRIPTION:
Cardiac surgery is associated with a significant risk of postoperative complications, including organ dysfunction such as acute kidney injury (AKI). Traditionally, clinical management in the intensive care unit (ICU) has focused on monitoring macrocirculatory parameters-such as blood pressure, cardiac output, and central venous pressure (CVP)-to guide treatment. However, adequate systemic perfusion does not always translate into sufficient tissue oxygenation at the microcirculatory level. Microcirculation, which occurs in the smallest vessels such as capillaries, is where oxygen and nutrients are actually delivered to the cells. Impairment in microcirculatory function can occur even when macrocirculatory values appear normal, leading to what is known as loss of hemodynamic coherence. Despite growing evidence of the clinical importance of microcirculation, routine bedside assessment remains limited due to technical challenges and the lack of easily applicable tools.

While elevated CVP and signs of venous congestion have been linked to worse outcomes such as AKI, the underlying mechanisms remain poorly understood. CVP alone is an imperfect marker for venous stasis and does not reliably predict microcirculatory impairment. Newer ultrasound-based tools-such as the Vexus score and femoral vein Doppler (FVD)-are emerging as promising, non-invasive methods to assess venous congestion at the bedside. However, it is currently unclear whether these sonographic signs of venous congestion are actually associated with impaired microcirculatory function. This knowledge gap limits clinicians' ability to interpret ultrasound findings in the context of microvascular health and to make informed decisions about fluid management and organ perfusion.

The VeMic study aims to investigate whether ultrasound-based indicators of venous congestion correlate with objectively measured microcirculatory impairment in patients admitted to the ICU after non-emergency cardiac surgery. By combining ultrasound assessments with advanced analysis of sublingual microcirculation using handheld vital microscopy and automated software, the study seeks to bridge the gap between macro- and microcirculatory monitoring. The findings may help determine whether these easily accessible ultrasound tools can be used to detect early signs of microvascular dysfunction and guide more targeted, physiology-based interventions in the postoperative setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective or urgent (need for definitive procedure during hospitalisation, but not emergency intervention) cardiac surgery

Exclusion Criteria:

* Age < 18 years
* Pregnant women
* Known severe chronic kidney disease (estimated glomerular filtration rate <15 mL/min per 1.73 m2 or dialysis)
* Renal or liver transplantation
* Any known condition interfering with Doppler evaluation of the portal system (including known or suspected cirrhosis or portal vein thrombosis or huge abdominal emphysema).
* Inability to consent to study
* Emergency cardiac surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting for elective or urgent cardiac surgery. Urgent patients are defined as patients who have not been electively admitted for operation but who require intervention or surgery on the current admission for medical reasons. These patients cannot be sent home without a definitive procedure but do not require immediate emergency surgery.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in red blood cell velocity: concested vs non-congested | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in red blood cell velocity (RBCv) between patients grouped as congested (Vexus score of 2 and 3) vs. non-congested (Vexus score of 0 and 1).
Difference in total vessel density: concested vs non-congested | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in total vessel density (TVD) between patients grouped as congested (Vexus score of 2 and 3) vs. non-congested (Vexus score of 0 and 1).
Difference in red blood cell velocity: physiologic femoral vein flow vs. pulsatile pattern | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in red blood cell velocity (RBCv) between patients with a physiologic femoral vein flow vs. pulsatile pattern
Difference in total vessel density between patients with a physiologic femoral vein flow vs. pulsatile pattern | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in total vessel density (TVD) between patients with a physiologic femoral vein flow vs. pulsatile pattern

SECONDARY OUTCOMES:
Difference in RBCv between patients with different Vexus scores | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in RBCv between patients with a Vexus score of 0 vs. 1 vs. 2 vs. 3
Difference inTVD between patients with different Vexus scores | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference inTVD between patients with a Vexus score of 0 vs. 1 vs. 2 vs. 3
Difference in microcirculatory reserve capacity: congested non-congested | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in microcirculatory reserve capacity between patients grouped as congested (Vexus score of 2 and 3) vs. non-congested (Vexus score of 0 and 1)
Difference in microcirculatory reserve capacity: physiologic femoral vein flow vs. pulsatile patern | 3 measurements:T0 prior surgery, T1 first post-operative day, T2 6 hours after T1
  Difference in microcirculatory reserve capacity between patients with a physiologic femoral vein flow vs. pulsatile patern

CONTACTS AND LOCATIONS:
Overall Officials: Martin Siegemund, Prof. MD, Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland